CLINICAL TRIAL: NCT03414242
Title: Investigation of Neurocognitive Measures of Sport-Related Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David B. Soma, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17-006025
Record Dates: First submitted 2018-01-10; First posted 2018-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Concussion, Brain
Keywords: brain; concussion; neck; strength; sport; prevention
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical spine musculature (Experimental)
  Interventions: Other: Cervical spine musculature

INTERVENTIONS:
Other: Cervical spine musculature — Previously established cervical spine musculature training methodology will be utilized to develop a concussion prevention training program.

SUMMARY:
The overall objective is to provide an onsite diagnosis with subsequent return to play criteria, as well as, lower the risk of traumatic brain injury by primary prevention through cervical spine neuromuscular control and vision training. The central hypothesis is that improved understanding of neurocognitive measures and function will provide improved diagnosis of concussion and help reduce the incidence of subsequent sports-related injury.

ELIGIBILITY:
Inclusion Criteria:

* 12-30 year old competitive or recreational athletes

Exclusion Criteria:

* Pre-existing condition preventing the ability to perform neck range of motion or a neck strength assessment
* Recent exposure to head lice
* Known or suspected pregnancy

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood metabolite profile | Through study completion, an athletic season average of 4 months
  Blood metabolite profile change from baseline blood draws will be analyzed to determine what blood biomarkers (e.g. amino acids, glycerophospholipids (mg/dL) ) are most sensitive to the presence of a concussion.

CONTACTS AND LOCATIONS:
Overall Officials: David Soma, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No